CLINICAL TRIAL: NCT06060418
Title: Effect of Lavender Aromatherapy on Post-Operative Nausea and Vomiting Among Laparotomy Patients At DHQ Sheikhupura Punjab, Pakistan
Brief Title: Effect of Lavender Aromatherapy on Post-Operative Nausea and Vomiting Among Laparotomy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Nosheen Siddique, MS Nursing Scholar, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aroma RCT 2023
Record Dates: First submitted 2023-09-18; First posted 2023-09-29 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: After deciding the participant of intervention group the researcher will start the protocol of intervention The intervention will start if NRS score is > 1 for nausea and with the 1st episode of vomiting.
  The researcher will soak a 4×4 cm sterile gauze pad with 0.2 ml equivalent to 2 drops of 10% Lavender essential oil and will suspended the soaked gauze at a distance of 10cm from the patient's nose with the help of forcep, and he or she will have asked to inhale its scent for 5 min. 15 and 40 minutes after the beginning of the aromatherapy treatment, the researcher will measure the nausea and vomiting scores by using the standardized tool. During this entire 40 minutes the researcher will strictly monitor the participant's condition. If the nausea score will be still higher than 1 or vomiting persists the participants will be noted as failure of treatment and move to standard care and the control group received standard care against the complain of nausea and vomiting.
Who Masked: Outcomes Assessor
Masking Description: The ward Manager/Head Nurse will act as an outcome assessor and blind to the intervention group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): After deciding on the participant of the intervention group the researcher will start the protocol of intervention The researcher will soak a 4×4 cm sterile gauze pad with 0.2 ml equivalent to 2 drops of 10% Lavender essential oil and will suspend the soaked gauze at a distance of 10cm from the patient's nose with the help of forceps, and he or she will have asked to inhale its scent for 5 min. 15 and 40 minutes after the beginning of the aromatherapy treatment, the researcher will measure the nausea and vomiting scores by using the standardized tool. During this entire 40 minutes, the researcher will strictly monitor the participant's condition. If the nausea score is still higher than 1 or the vomiting persists the participants will be noted as failure of treatment and move to standard care.
  Interventions: Other: aromtherapy
- Control group (No Intervention): The control group received standard care against the complain of nausea and vomiting.

INTERVENTIONS:
Other: aromtherapy — aromatherapy with essential oil is being used as a non-pharmacological nursing intervention within the health care setting. This approach aims to manage the patient's discomfort and alleviate the symptoms of postoperative nausea and vomiting. One of the most beneficial oils is Lavender Essential Oil (LEO), which is used to treat a variety of digestive issues.
  Arms: Intervention Group

SUMMARY:
Post-operative nausea and vomiting are critical problems that occur commonly after the administration of general anesthesia, which can lead to serious health complications such as hemorrhage, electrolyte imbalance and ultimate shock. To prevent these complications, antiemetic drugs are often administered, but they can cause side effects as well as increased healthcare costs. As concerns regarding the side effects of antiemetic drugs have grown, there has been an increased interest in using non-pharmacologic interventions, such as aromatherapy, as an alternative approach to preventing post-operative nausea and vomiting. It involves the therapeutic use of essential oils, and lavender essential oil, in particular, is commonly used for various digestive problems including nausea, and vomiting. Therefore, a key question for a health care professional is how to prevent post-operative nausea and vomiting in best possible manner? To address this question, a study will be conducted in District Head Quarter Sheikhupura, aiming to evaluate the effectiveness of lavender essential oil aromatherapy in reducing post-operative nausea and vomiting among patients admitted for laparotomy under general anesthesia. This study will be a Randomized control trial with the study population consisting of admitted patients after laparotomy under general anesthesia. The sample size will be 70, who will be divided into two groups, each consisting of 35 participants. A convenience sampling technique will be employed for the recruitment of participants. After that, the participants will be randomized into control and intervention groups by computer-generated table numbers in accordance with the inclusion criteria that is, 18-65 age, both genders, laparotomy under general anesthesia, clinically stable, and susceptive to post-op nausea and vomiting within 24hrs following the surgery. whereas, the patients with respiratory diseases, allergies, infections, reversal laparotomy within short duration, having any kind of addiction, those who move to the intensive care unit, those with a history of motion sickness, history of pre-op nausea and vomiting and those who start oral or NG feed before 24hrs will not be part of this study. The data will be analyzed by using Statistical Package for Social Sciences version 22.

DETAILED DESCRIPTION:
Study Design:

Randomized Control trial( RCT)

Study population:

Patients undergoing laparotomy under general anesthesia

Setting:

This study will be carried out at the Institute of Nursing, University of Health Sciences Lahore in collaboration with DHQ Sheikhupura Punjab, Pakistan. This hospital offers 24/7 services in emergency, medicine, surgery, gynecology and pediatrics etc.

Sample Size:

The sample size for each group is 35 and total is 70.

Sampling Technique and Randomization:

A non-probability convenience sampling approach will be utilized for patient enrollment. patients will be randomly assigned to either the intervention or control group through computer-generated table numbers.

Data Collection Procedure and Method of Intervention; Upon receiving approval from the Institutional Review Board of the University of Health Sciences Lahore, formal authorization will be sought from DHQ. Eligible participants will be identified and selected in accordance with predetermined inclusion and exclusion criteria. After explaining the study purpose, the researcher will obtain informed written consent before their surgical procedure. Upon patients' arrival to the HDU following their laparotomy, those who present complaints of postoperative nausea and vomiting will be subject to randomization into either the intervention or control group. This randomization will be executed using computer-generated table numbers. First, the researcher will gather pertinent demographic information from the enrolled participants.

Adequate guarantees of confidentiality shall be extended to all participants.

Method of Intervention:

After deciding the participant of intervention group the intervention will be started if NRS score is > 1 for nausea and with the 1st episode of vomiting.

The researcher will soak a 4×4 cm sterile gauze pad with 0.2 ml equivalent to 2 drops of 10% Lavender essential oil and will suspended the soaked gauze at a distance of 10cm from the patient's nose with the help of forcep, and he or she will have asked to inhale its scent for 5 min. 15 and 40 minutes after the beginning of the aromatherapy treatment, the researcher will measure the nausea and vomiting scores by using the standardized tool. During this entire 40 minutes the researcher will strictly monitor the participant's condition. If the nausea score will be still higher than 1 or vomiting persists the participants will be noted as failure of treatment and move to standard care and the control group received standard care against the complaint of nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

Those patients: -

* with 18 -65 years
* both Male and Female
* who received general anesthesia for surgery
* who experience nausea and vomiting within 24hr after surgery
* who hemodynamically stable

Exclusion Criteria:

Those patients

* • who move to ICU after the Procedure

  * with history of substance addiction
  * having history of pre-op nausea and vomiting
  * with history of motion sickness
  * who start Oral or Naso Gastric Feed after surgery
  * having history of Lung disease, ant type of allergy or infection
  * who need laparotomy reversal short after the procedure
  * Who received antiemetic before surgery
  * who went to any type of complication during the procedure not included in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of postoperative nausea Intensity | with in 24 hour after the surgery
  When a patient encounters nausea within the initial 24 hours subsequent to the laparotomy, the researcher will adopt the Numeric Rating Scale (NRS) to quantify the intensity of the experienced nausea.
  The NRS is a one-dimensional quantitative 11-point pain rating scale that has also been validated to detect nausea by using the content validity method, and its score is 1 which is appropriate to measure the nausea intensity. The researcher will operate this scale by using the verbal scale because self-assessed nausea scores from the NRS and the verbal scale correlated well as rSpearman = 0.79. The researcher will ask the patient to select a number from 0 to 10 that best describes the intensity of their nausea at that precise moment.
Measurement of postoperative Vomiting frequency and severity | with in 24 hour after the surgery
  in scenarios where a patient reports episodes of vomiting during the initial 24-hour postoperative period, the researcher will utilize the Likert scale to assess both the frequency and severity of these vomiting incidents.
  Vomiting will be assessed by using a Likert Scale that was also validated on 10% of the sample size. The CVI was 1 and Cronbach alpha was 0.79 which is appropriate to measure the severity of vomiting. The researcher will rate the severity of vomiting as 0 to 4, with 0 representing no vomiting and 4 representing severe vomiting. The number of occurrences indicates the severity (0 = no episode, 1 = 1-2 episodes, 2 = 3-4 episodes, 3 = 5 or more episodes)

CONTACTS AND LOCATIONS:
Overall Officials: Nosheen Siddique, MSN, Principal Investigator — University of Health Sciences Lahore
Locations (1):
- Nosheen Siddique, Sheikhupura, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to share the data with other researchers after the analysis of the results. This will help the researchers to identify the gaps and further research covers the limitation of this study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After Publication the data will be available for other researchers.
Access Criteria: The criteria will be uploaded after the publication of this research